CLINICAL TRIAL: NCT06917872
Title: An Open-label, Fixed-sequence, Two-period Phase I Trial to Evaluate the Effect of Multiple Oral Doses of Erythromycin, a Moderate CYP3A4 Inhibitor, on the Pharmacokinetics of BI 1291583 at Steady State in Healthy Male and Female Subjects
Brief Title: A Study in Healthy People to Test Whether Erythromycin Influences the Amount of BI 1291583 in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1397-0029; 2024-515795-12-00 (Registry Identifier: CTIS); U1111-1310-2268 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2025-04-07; First posted 2025-04-09 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Healthy
MeSH Terms: interventions — Erythromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BI 1291583 alone followed by BI 1291583 + erythromycin (Experimental): Period 1 + period 2
  Interventions: Drug: BI 1291583; Drug: erythromycin

INTERVENTIONS:
Drug: BI 1291583 — BI 1291583
  Other Names: Verducatib
Drug: erythromycin — erythromycin

SUMMARY:
The main objective of this trial is to investigate the effect of erythromycin, a moderate CYP3A4 inhibitor on the pharmacokinetics of BI 1291583 at steady state.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 50 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent in accordance with ICH Harmonized Guideline for Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial
* Male subject, willing to use male contraception (condom or sexual abstinence) and to refrain from sperm donation from time point of administration of trial medication until 90 days after last administration of trial medication, if their sexual partner is a woman of child-bearing potential (WOCBP) or

Female subject who meets any of the following criteria for a highly effective contraception from at least 30 days prior to first administration of trial medication until 5 months after last administration of trial medication:

* Use of combined (estrogen and progestogen containing) hormonal contraception that prevents ovulation (oral, intravaginal or transdermal), plus condom in male partner
* Use of progestogen-only hormonal contraception that inhibits ovulation (only injectables or implants), plus condom in male partner
* Use of intrauterine device (IUD) or intrauterine hormone-releasing system (IUS), plus condom in male partner
* Sexually abstinent
* Male sexual partner of the trial participant is vasectomized and received medical assessment of the surgical success of the vasectomy (documented absence of sperm)
* Surgically sterilized (including hysterectomy, bilateral salpingectomy, bilateral oophorectomy, or bilateral tubal occlusion)
* Postmenopausal, defined as no menses for 1 year without an alternative medical cause (in questionable cases a blood sample with levels of follicle-stimulating hormone (FSH) above 40 U/L and estradiol below 30 ng/L is confirmatory)

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the Investigator
* Repeated measurement of systolic BP outside the range of 90 to 140 mmHg, diastolic BP outside the range of 50 to 90 mmHg, or PR outside the range of 50 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance (including but not limited to electrolyte disturbances, particularly hypokalemia and hypomagnesemia)
* Any evidence of a concomitant disease assessed as clinically relevant by the Investigator
* Any known gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, hormonal or immunological disorders (including any known relevant immunodeficiency)
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2025-04-29 (Actual); Primary Completion 2025-09-09 (Actual); Study Completion 2025-09-09 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of BI 1291583 in plasma at steady state over a uniform dosing interval τ (AUCτ,ss) | Up to 72 days
Maximum measured concentration of BI 1291583 in plasma at steady state over a uniform dosing interval τ (Cmax,ss) | Up to 72 days

SECONDARY OUTCOMES:
Time from last dosing to maximum concentration of BI 1291583 in plasma at steady state (tmax,ss) | Up to 72 days
Minimum concentration of BI 1291583 in plasma at steady state within a uniform dosing interval τ (Cmin,ss) | Up to 72 days

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Berlin GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com